CLINICAL TRIAL: NCT02398175
Title: Thoracic Injuries in Pediatric Polytraumatized Patients: Epidemiology, Treatment and Outcome
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 2008
Record Dates: First submitted 2015-03-16; First posted 2015-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Trauma
Keywords: Pediatric polytrauma; thoracic injuries
MeSH Terms: conditions — Multiple Trauma; Thoracic Injuries | interventions — Resuscitation; Intubation

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Pediatric polytraumatized patients with thoracic injuries: Pediatric polytraumatized patients (age < 18), (ISS > 16) with thoracic injuries
  Interventions: Other: reanimation/intubation

INTERVENTIONS:
Other: reanimation/intubation

SUMMARY:
The present study predicts that concomitant chest injuries in polytraumatized pediatric patients are a potential source of substantial morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

Children with isolated, but severe and potentially life-threatening injuries ISS ≥16 injuries to only one body cavity together with a single long bone fracture thoracic injuries

Exclusion Criteria:

Injury Severity Score (ISS) of < 16 age >18 no thoracic injuries

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric (age < 18 years) polytrauma patients with associated thoracic injuries, admitted to this Level I Trauma center, between January 1992 and December 2008
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2008-01; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Injury Severity Score | at least one year follow up
Thoracic Injuries | at least one year follow up
  Thoracic injuries and outcome ( number of participants with Thoracic Injuries, type of injury)